CLINICAL TRIAL: NCT03869619
Title: REAL WORLD DATA IN LYMPHOMA AND SURVIVAL IN ADULTS
Acronym: REALYSA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0352; 2018-A01332-53 (Other: ID-RCB)
Record Dates: First submitted 2018-08-16; First posted 2019-03-11 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Diffuse Large B Lymphoma (DLBCL); Follicular Lymphoma (FL); Mantle Cell Lymphoma (MCL); Marginal Zone Lymphoma (MZL); T-cell Lymphoma (T-NHL); Hodgkin's Lymphoma (HL); Burkitt Lymphoma (BL))
Keywords: lymphoma; real life; cohort; epidemiology; PRO
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell; Hodgkin Disease; Burkitt Lymphoma; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All enrolled patients: All patient who signed the consent form for participation to the study
  Interventions: Other: Real-life epidemiological platform of lymphoma in France

INTERVENTIONS:
Other: Real-life epidemiological platform of lymphoma in France — The REALYSA database will be described with the following characteristics:
  * Number of patients included per month in total and according to subtype of lymphoma
  * Number of patients in each region in total and according to subtype of lymphoma

SUMMARY:
REALYSA cohort is a population-based epidemiological platform in real-life for lymphomas designed to enrich prognostic data, by integrating together epidemiological, clinical and biological data.

REALYSA is a platform perfectly set up to

* Study prognostic factors using integrated epidemiological and biological data (genetics), to better characterize the determinants of refractoriness and relapse in patients with lymphoma, to follow the growing number of survivors and describe median to long-term sequela, second cancer, quality of life (QoL)…
* Document treatment effectiveness in real life and observance
* Address socio-economical questions

ELIGIBILITY:
Inclusion Criteria:

* Signature of the consent form for participation in the REALYSA cohort
* Aged over 18 at the time of inclusion
* Diagnosed with lymphoma in the last 6 months (180 days)
* Lymphoma subtype belonging to at least one of the 7 histological subtypes: diffuse large B-cell lymphoma, follicular lymphoma, mantle cell lymphoma, marginal zone lymphoma, T-cell lymphoma, Hodgkin's lymphoma, Burkitt lymphoma

Exclusion Criteria:

* Anti-lymphoma treatment already received (except pre-phase: typically corticosteroids, vincristine, cyclophosphamide, etoposide, alone or in combination)
* Documented HIV infection
* Any other lymphoma subtype not included in the list in Appendix 1. Of note, are excluded:

  * Chronic lymphocytic leukemia/small lymphocytic lymphoma
  * Hairy cell leukemia and variant
  * Lymphoplasmacytic lymphoma
  * Waldenström macroglobulinemia
  * Primary DLBCL of the central nervous system (CNS)
  * T-cell large granular lymphocytic leukemia
  * Chronic lymphoproliferative disorder of NK cells
  * Mycosis fungoides
  * Sézary syndrome
  * Primary cutaneous T cell lymphomas (mainly diagnosed and treated by dermatologists)
  * Post-transplant lymphoproliferative disorders (PTLD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with lymphoma in the last 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2027-11-14 (Estimated); Study Completion 2027-11-14 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 5 years

SECONDARY OUTCOMES:
Number of patients included per month in total and according to subtype of lymphoma | 5 years
Number of patients in each region in total and according to subtype of lymphoma | 9 years
Progression-Free Survival (PFS) | 9 years
Event-Free Survival (EFS) | 5 years
Event-Free Survival (EFS) | 9 years
Overall Survival (OS) | 5 years
Overall Survival (OS) | 9 years
Net Survival | 5 years
Net Survival | 9 years
Response rate | 5 years
Response rate | 9 years
Duration of response | 5 years
Duration of response | 9 years
Time to Next Anti-Lymphoma Treatment (TTNLT) | 5 years
Time to Next Anti-Lymphoma Treatment (TTNLT) | 9 years
Duration of Survival after progression | 5 years
Duration of Survival after progression | 9 years
Frequency of Lymphoma transformations | 5 years
Frequency of Lymphoma transformations | 9 years
Frequency of Second cancers | 5 years
Frequency of Second cancers | 9 years
Frequency of other chronic disease | 5 years
Frequency of other chronic disease | 9 years
Number of exposure factors | Baseline
Number of comorbidities | Baseline

OTHER OUTCOMES:
Representativeness of the included population | 5 years
  Study population must show a good representativeness of the source population regarding demographic or diseases characteristics, to be able to generalize our results. Indeed, the representativeness of the study population can only be evaluated in areas covered by population-based cancer registries (PBCR) by comparing cases included in the REALYSA project to incident lymphoma cases registered in the general population (PBCR of the FRANCIM network).
Representativeness of the included population | 9 years
  Study population must show a good representativeness of the source population regarding demographic or diseases characteristics, to be able to generalize our results. Indeed, the representativeness of the study population can only be evaluated in areas covered by population-based cancer registries (PBCR) by comparing cases included in the REALYSA project to incident lymphoma cases registered in the general population (PBCR of the FRANCIM network).

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Ghesquières, MD, Study Director — Hospices Civils de Lyon; Alain Monnereau, MD, Study Director — Université de Bordeaux : Inserm
Locations (37):
- France (37):
  - Unité d'Hématologie Clinique, CH D'ARRAS, Arras
  - Service d'Hématologie, CHU Jean Minjoz, Besançon
  - Service d'Onco-radiolothérapie, Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - Service d'Hématologie, Institut d'Hématologie de Basse Normandie, Caen
  - METROPOLE SAVOIE - SITE CHAMBERY, place Lucien Biset,, Chambéry
  - Service d'Hématologie Clinique et de Thérapie Cellulaire, Hôpital Estaing, CHU de Clermont-Ferrand, Clermont-Ferrand
  - Unité Hémopathies Lymphoïdes, Hôpital Henri Mondor, Créteil
  - CHU Francois MITTERRAND, Dijon
  - Service Hématologie, Centre Hospitalier de Dunkerque, Dunkirk
  - Service Oncologie médicale, Groupe Hospitalier Mutualiste de Grenoble, Institut Daniel Hollard,, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Service d'Hématologie Clinique, Centre Hospitalier Universitaire Michallon, La Tronche
  - Clinique Victor Hugo, Le Mans
  - Centre hospitalier Libourne, Libourne
  - Service Oncologie médicale, HOPITAL SAINT VINCENT-DE-PAUL, Lille
  - Service des maladies du sang, Hôpital Claude Huriez, CHRU de Lille, Lille
  - Service Hématologie Clinique et Thérapie Cellulaire, CHU DE LIMOGES - HOPITAL DUPUYTREN,, Limoges
  - Département d'Hématologie et Oncologie, Centre Léon Bérard, Lyon
  - Département d'Hématologie Clinique, Hôpital Saint-Eloi,, Montpellier
  - Service Hématologie, GH REGION MULHOUSE ET SUD ALSACE - HOPITAL EMILE MULLER,, Mulhouse
  - Service d'Hématologie clinique, Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier de Niort, Niort
  - Service Hématologie, Hôpital St Louis, Paris
  - CHU Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Service d'Hématologie et Thérapie Cellulaire, Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hématologie Clinique, CHU PONTCHAILLOU, Rennes
  - Service Hématologie, Centre Hospitalier de Roubaix - Hôpital Victor Provo, Roubaix
  - Service Hématologie, UNIVERSITE DE ROUEN, CENTRE HENRI BECQUEREL, Rouen
  - Service Hématologie, CH YVES LE FOLL, Saint-Brieuc
  - Service Hématologie, Institut Curie - Hôpital René HUGUENIN, Saint-Cloud
  - Département d'Hématologie Clinique et Thérapie Cellulaire, Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer, Toulouse
  - Hématologie Clinique, CH DE BRETAGNE ATLANTIQUE, Vannes

REFERENCES:
- [Derived] Ghesquieres H, Cherblanc F, Belot A, Micon S, Bouabdallah KK, Esnault C, Fornecker LM, Thokagevistk K, Bonjour M, Bijou F, Haioun C, Morineau N, Ysebaert L, Damaj G, Tessoulin B, Guidez S, Morschhauser F, Thieblemont C, Chauchet A, Gressin R, Jardin F, Fruchart C, Laboure G, Fouillet L, Lionne-Huyghe P, Bonnet A, Lebras L, Amorim S, Leyronnas C, Olivier G, Guieze R, Houot R, Launay V, Drenou B, Fitoussi O, Detourmignies L, Abraham J, Soussain C, Lachenal F, Pica GM, Fogarty P, Cony-Makhoul P, Bernier A, Le Guyader-Peyrou S, Monnereau A, Boissard F, Rossi C, Camus V. Challenges for quality and utilization of real-world data for diffuse large B-cell lymphoma in REALYSA, a LYSA cohort. Blood Adv. 2024 Jan 23;8(2):296-308. doi: 10.1182/bloodadvances.2023010798. PMID 37874913
- [Derived] Ghesquieres H, Rossi C, Cherblanc F, Le Guyader-Peyrou S, Bijou F, Sujobert P, Fabbro-Peray P, Bernier A, Belot A, Chartier L, Fornecker LM, Baldi I, Bouabdallah K, Laurent C, Oberic L, Morineau N, Le Gouill S, Morschhauser F, Haioun C, Damaj G, Guidez S, Laboure G, Fitoussi O, Lebras L, Gressin R, Salles G, Ysebaert L, Monnereau A. A French multicentric prospective prognostic cohort with epidemiological, clinical, biological and treatment information to improve knowledge on lymphoma patients: study protocol of the "REal world dAta in LYmphoma and survival in adults" (REALYSA) cohort. BMC Public Health. 2021 Mar 2;21(1):432. doi: 10.1186/s12889-021-10433-4. PMID 33653294